CLINICAL TRIAL: NCT02685228
Title: Clinical Study of Low Dose of Decitabine Combined With Gemcitabine in First-line Treatment of Locally Advanced, Unresectable or Metastatic Pancreatic Cancer
Brief Title: Decitabine Combined With Gemcitabine in First-line Treatment of AdvancedPancreatic Cancer
Acronym: SLOWDOSE001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLOWDOSE001
Record Dates: First submitted 2016-02-01; First posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Decitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- decitabine & gemcitabine (Experimental): This group was treated by low dose decitabine combinated with gemcitabine regimen. decitabine: 5mg/m2 d1-d5; gemcitabine: 1.0g/m2,d8,d15,d22. 28days for one cycle.
  every 28days for one cycle
  Interventions: Drug: Decitabine; Drug: Gemcitabine
- gemcitabine (Active Comparator): This group was treated by gemcitabine only. Gemcitabine: 1.0g/m2, d8,d15,d22; 28 days for one cycle. every 28days for one cycle
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Decitabine — decitabine 5mg/m2,d1-d5;
  Arms: decitabine & gemcitabine
Drug: Gemcitabine — gemcitabine 1.0g/m2, d8,d15,d22

SUMMARY:
The purpose of this study is to investigate the effect of very low dose decitabine combinate with gemcitabine in the first-line treatment of locally advanced, unresectable and metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This study intends to advanced pancreatic cancer with row standard with district group random way is divided into two groups, a group for the gemcitabine monotherapy in the treatment group, another group of gemcitabine combined with low dose of decitabine treatment group. The overall survival, progression free survival, and disease control rate were observed in patients treated with combined therapy. At the same time, its safety and tolerance were observed. The methylation status and its influence on the immune function were also detected by biological test.

ELIGIBILITY:
Inclusion Criteria:

* histology or cytology proved to be a local development, non excision or metastatic pancreatic cancer patients. Or clinical compliance, but the pathological specimens were difficult, can be fully communicated with patients, selected clinical research.
* in the treatment of advanced cancer with no anti tumor drug.
* the damage had been recovered by other treatments, in which patients received surgery for more than 2 weeks.
* aged 18-70 years
* the physical condition ECOG score (PS) is 0-1
* the expected survival time is greater than or equal to 12 weeks
* according to RECIST standard 1.1 there is at least one measurable lesion, and the lesion is irradiated with at least one measurable lesion. Any of the following methods can accurately measure the diameter of the lesions, the abdominal computed tomography CT or MRI, the conventional method of diameter of at least 20mm or the application of spiral CT diameter at least 10mm.
* the main organ function is normal, that is, in line with the following standards:(1) blood examination standard should meet: HB than 90g/L (without blood transfusion within 14 days), ANC = 1.5 * 109/L; PLT = 100 * 109/L.(2) biochemical examination must meet the following criteria: serum bilirubin is less than or equal to 1.5 times the upper limit of normal value, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) is less than or equal to 2.5 times the upper limit of the normal value of (if have hepatic metastasis allows ast, ALT is less than or equal to five times the upper limit of normal value). Serum creatinine was 1.5 times the upper limit of the normal value; creatinine clearance rate was 50mL/min.
* women of childbearing age must have a pregnancy test (serum or urine) within 7 days of entry, and the results are negative, and are willing to use appropriate methods of contraception within 8 weeks of the trial period and the last administered drugs. For men, must be agreed during the test and 8 weeks after administration of the test drug use contraceptive methods or surgical sterilization is appropriate.
* patients with good compliance.
* patients understand and voluntarily sign written informed consent.

Exclusion Criteria:

* the current or previous diagnosis of pancreatic cancer had no systemic anticancer therapy, including cytotoxic drug therapy, target to drug treatment, test treatment, auxiliary chemotherapy or neoadjuvant chemotherapy patients (but stopping for more than 6 months postoperative recurrence patients can be selected).
* patients with no measurable lesions, such as malignant pleural effusion and ascites, lymph node metastasis, bone metastasis, and brain spinal cord membrane.
* any effect on the patient's intravenous injection, and any effect on the absorption of the drug or the pharmacokinetic parameters of the drug.
* patients with systemic disease (such as unstable or non compensatory respiratory, cardiac, liver or kidney disease) with severe or no control. Any unstable systemic disease (including active infection, grade four hypertension, unstable angina, congestive heart failure, liver and kidney, or metabolic disease). Any other malignant tumor in the five years (except for the complete cure of cervical carcinoma in situ or basal cell or squamous cell skin cancer). There is a history of clear neurological or mental disorders, including epilepsy or dementia.
* patients with the functional level of the various organs of the functional level of the existence of any other important clinical abnormalities or laboratory results so that patients do not fit to participate in the study of evidence. According to the National Cancer Institute common chemotherapy toxicity grading standards (NCI-CTC, 4 edition) has more than 2 levels of chronic toxicity (not including hair loss) not cured.
* known any severe allergic components of decitabine, gemcitabine.
* previous studies have been registered for the treatment of this study, or from the patients in this study were unable to enter the group.
* pregnancy or lactation women. 9) the researchers believe that the subjects may not be able to complete the study or may not be able to comply with the requirements of this study (as a result of management reasons or other reasons).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 24 months

SECONDARY OUTCOMES:
Evidence of the size of the lesion in pancreas confirmed by non-investigational CT or MRI | within every 28 days(plus or minus 3 days) ,up to 36 days. From date of randomization until the date of death from any cause, assessed up to 50 months.

IPD SHARING:
Plan to Share IPD: No